CLINICAL TRIAL: NCT02980614
Title: Cardiac 4D MR Velocity Mapping in Repaired Tetralogy of Fallot Patients: Evaluation of Pulmonary Regurgitant Fraction and Ventricular Volume
Brief Title: 4D Velocity Mapping of the Heart in rTOF Patients
Acronym: CARDIOFLUX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2016_843_0026
Record Dates: First submitted 2016-11-10; First posted 2016-12-02 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Magnetic Resonance Imaging; Tetralogy of Fallot
Keywords: phase-contrast MRI; blood flow; velocity mapping; Quantitative MRI; Cardiac imaging; Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants to 4D flow imaging (Experimental): In addition to the standard clinical MR protocol, 2 added sequences:
  4D MR sequence in cine mode 4D velocity mapping sequence
  Interventions: Device: 4D flow imaging

INTERVENTIONS:
Device: 4D flow imaging — To compare the quantification of pulmonary valve leakage by standard 2D flow MRI and 4D flow MRI by measuring the regurgitation fraction (ratio of retrograde blood flow to anterograde flow) in the pulmonary artery

SUMMARY:
MRI with 4D flow permits to assess the hemodynamic parameters in a parent vessel and its branches inside the same sequence.

DETAILED DESCRIPTION:
MRI with 4D flow permits to assess the hemodynamic parameters in a parent vessel and its branches inside the same sequence. The objective of the project is to compare the regurgitant fraction in the pulmonary artery (PA) measured using 4D MR-flow and standard 2D MR-flow in repaired Tetralogy of Fallot (rTOF) patients. The consistency of the 4D flow quantization will be assessed assuming mass conservation in the pulmonary artery tree (PA flow =LeftPA flow +RightPA flow ? ).

ELIGIBILITY:
Inclusion Criteria:

* Tetralogy of Fallot patients
* referred for clinical MRI examination
* ≥ 15 years

Exclusion Criteria:

* Anyone with a classic contraindication to MRI
* Severe obesity
* Gadolinium chelate allergy
* < 15 years
* counter-indication to MRI examination
* vulnerable person

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Regurgitant fraction comparison | Day 0
  The primary objective of the project is to compare the regurgitant fraction in the pulmonary artery (PA) measured with 4D MR-flow and standard 2D MR-flow.

SECONDARY OUTCOMES:
Right ventricular volume | Day 0
  The secondary objective is to compare the right ventricular volumes measured using the 4D prototype and the standard steady-state free precession sequences.
Pulmonary arteries flows | Day 0
  The consistency of the 4D flow quantization will be assessed assuming mass conservation in the pulmonary artery (PA) tree (PA flow =LeftPA flow +RightPA flow ? ).

CONTACTS AND LOCATIONS:
Overall Officials: Cedric Renard, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No